CLINICAL TRIAL: NCT03189199
Title: A Registry Study on Safety Surveillance of Dazhuhongjingtian (a Chinese Medicine
Brief Title: A Registry Study on Safety Surveillance of Dazhuhongjingtian (a Chinese Medicine Injection) Used in China
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: China Academy of Chinese Medical Sciences (Other)
Collaborators: Hospital of Changchun University of Traditional Chinese Medicine (Unknown)
Responsible Party: Principal Investigator, Yanming Xie, Deputy Director, China Academy of Chinese Medical Sciences
Other Study IDs: RSCMI-12
Record Dates: First submitted 2017-06-14; First posted 2017-06-16 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: a cohort using Dazhuhongjingtian injection — All patients will be measured and assessed at the time Dazhuhongjingtian Injection is administered to them until they discharge. Patients using Dazhuhongjingtian Injection will be registered on a registration form including disease background, Dazhuhongjingtian Injection's administration, and extraction information from hospital information system. An adverse event or drug adverse reaction form also will be used to describe any doubted symptoms or signs from patients. A judgment will be made by doctors directly and a further analysis will be conducted by researchers to decide those potential side effects of Dazhuhongjingtian Injection.

SUMMARY:
The purpose of this study is to make a cohort event monitoring to see whether and how Dazhuhongjingtian injection in hospital results in adverse events or adverse drug reactions

DETAILED DESCRIPTION:
Safety surveillance on Chinese Medicine injection is an important problem that needs to be sorted out ,because in mainland China hospitals ,Chinese Medicine Injection are used widely. Population for taking medicine characteristics,the incidence rate of ADR and other uncertain factors influence can few be found now.A registry study for Dazhuhongjingtian injection safety surveillance with 3000 patients will be conducted from June.2017 to Dec.2019.Eligibility criteria Patients who will use Dazhuhongjingtian injection in 4 selected hospitals from2017-2019.

ELIGIBILITY:
Inclusion Criteria:

- An anticipated sample size was caculated in this study, about 3000. Patients using Dazhuhongjingtian injection from 2017 to 2019 in 4 hospitals

Exclusion Criteria:

none

Min Age: 1 Hour | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: An anticipated sample size was caculated in this study, about 3000. Patients using Dazhuhongjingtian injection from 2017 to 2019 in 4 hospitals
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2017-06-19 (Estimated); Primary Completion 2017-07-19 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dazhuhongjingtian's ADRs,especially number of participants with adverse events. | The registry procedure will last about 3 years only for patients using Dazhuhongjingtian
  All patients will be measured and assessed at the time Dazhuhongjingtian is administered to them until they discharge. Patients using Dazhuhongjingtian will be registered on a registration form including disease background, Dazhuhongjingtian's administration, and extraction information from hospital information system. An adverse event or drug adverse reaction form also will be used to describe any doubted symptoms or signs from patients. A judgment will be made by doctors directly and a further analysis will be conducted by researchers to decide those potential side effects of Dazhuhongjingtian.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Ming Xie, BA, Study Chair — Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences

IPD SHARING:
Plan to Share IPD: Yes